CLINICAL TRIAL: NCT05342688
Title: Associations Between Contextual Interference, Engagement During Treatment, and Change in Motor Performance Among Patients Posts-stroke
Brief Title: Contextual Interference, Engagement , and Change in Motor Performance in Stroke
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Collaborators: Reuth Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Michal Kafri, PhD, Principal Investigator, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0012-19-RRH
Record Dates: First submitted 2021-11-09; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Hemiparesis;Poststroke/CVA

STUDY DESIGN:
Intervention Model Description: The study will be a randomized controlled trial with a pre-post design.
Who Masked: Outcomes Assessor
Masking Description: Masking description: The outcome assessor will be blind to the group assignment of the participants. Participants and the investigator who deliver the intervention will be aware of group assignment because it is inherent to the type of practice they receive and deliver respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High contextual interference (Experimental): The intervention will involve practicing three items from the Wolf motor function test in random order during three sessions. Each item will be repeated 30 times in total.
  Interventions: Behavioral: Task-specific practice of upper extremity functions
- Low contextual interference (Active Comparator): The intervention will involve practicing three items from the Wolf motor function test in blocked order during three sessions. Each item will be repeated 30 times in total.
  Interventions: Behavioral: Task-specific practice of upper extremity functions

INTERVENTIONS:
Behavioral: Task-specific practice of upper extremity functions — The intervention will consist of training of items from the Wolf motor function test.

SUMMARY:
The aim of the study is to examine associations between contextual interference (CI), engagement during practice and changes in upper limb motor performance among patients post-stroke.

Fifty patients over the age of 18, after a stroke, in the sub-acute and early chronic stages who have weakness of the upper extremity and are treated in a rehabilitation center will be recruited.

The study will include participation in five sessions: session 1 for baseline assessment, session 2-4 for practice of upper extremity functions, and session 5 for post intervention assessment. The intervention will include training of three items from the Wolf motor function test in random order (high CI group) or block order (low CI group). Outcomes of engagement will include the brain engagement index, heart rate variability and galvanic skin response. Outcomes of learning will include the pre-post change in performance of the wolf motor function selected items.

DETAILED DESCRIPTION:
The aim of the study is to examine associations between contextual interference (CI), engagement during practice, and changes in upper limb motor performance among patients post-stroke.

Fifty patients over the age of 18, after a stroke, in the sub-acute and early chronic stages who are treated in a rehabilitation center inpatient or outpatient clinics, who have hemiparesis (Fugl-Meyer score = 11-60) will be recruited.

Patients with a history of neurological diseases other than stroke or orthopedics conditions that impair upper extremity function, pain that prevents active movement, hemodynamic instability, cognitive decline and language difficulties that do not allow understanding of instructions and cooperation will be excluded.

The study will include participation in five sessions. In the first session, participants will answer a demographic questionnaire and a set of motor (including the Wolf motor function test), perception and cognitive tests will be delivered. Then participants will be assigned to either high or low CI groups. In the next three sessions, participants will practice three items from the Wolf motor functions test. Participants in the high CI group will practice the items in random order and those in the low CI group will practice the selected items in blocked order. Assessment of outcomes during practice will include assessment of brain engagement index by recording EEG (one electrode) and heart rate variability and galvanic skin response. In the fifth session, at the end of the intervention, a reassessment of the wolf motor function performance will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Five days to 1-year post-stroke
* Score of 11-60 on the Fugl-Meyer Assessment for upper extremity
* The patient receives physical therapy and/or occupational therapy rehabilitation treatment

Exclusion Criteria:

* A history of neurological diseases other than stroke or orthopedics conditions that impair upper extremity function
* Pain that prevents active movement of the upper extremity
* Hemodynamic instability
* Cognitive decline and language difficulties that do not allow understanding of instructions and cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in Brain Engagement Index | Practice session 1 (1-2 days following pre-intervention session), practice session 2 (1-2 days following practice session1), and practice session 3 (1-2 days following practice session1)
  EEG activity in the prefrontal cortex will be measured by MindWave mobile EEG headset.
Change in time to complete each of three items of the Wolf Motor Function Test (WMFT) | Pre-intervention session (first session), post-intervention session (session 5, 5-7 days following the pre-intervention session))
  A maximum of 120 seconds is allowed. Any performance that exceeds 120 seconds is assigned 120 seconds.

SECONDARY OUTCOMES:
Changes in Heart rate variability | Practice session 1 (1-2 days following pre-intervention session), practice session 2 (1-2 days following practice session1), and practice session 3 (1-2 days following practice session1)
  Photoplethysmograph sensor will be placed on the ring finger. Data will be used to extract R-R beat interval, and variability will be measured.
Changes in Galvanic Skin Response (GSR) | Practice session 1 (1-2 days following pre-intervention session), practice session 2 (1-2 days following practice session1), and practice session 3 (1-2 days following practice session1)
  GSR electrodes will be placed on the index and middle fingers, and the signal is reported in micro-Siemens (μS) units.

CONTACTS AND LOCATIONS:
Locations (1):
- Reut Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No